CLINICAL TRIAL: NCT01207635
Title: Evaluation of Antiproliferative Effects of Arimidex in Ductal Lavage Fluid in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LAB02-0400
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Cancer; Arimidex
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood drawn; and, fluids collected from ductal lavage.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Patients
  Interventions: Procedure: Ductal Lavage Fluid Collection

INTERVENTIONS:
Procedure: Ductal Lavage Fluid Collection — Procedure of inserting a small catheter into the ductal openings in the nipple and washing out cells from inside the duct.

SUMMARY:
The goal of this study is to evaluate antiproliferative effects of Arimidex in ductal lavage fluids of Breast Cancer patients.

Breast cancer is the leading cause of cancer incidence and the second leading cause of cancer mortality in women. Breast duct fluid provide biomarkers to aid in risk assessment of developing breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a history of breast cancer.
* Patient must be scheduled to receive standard treatment with Arimidex for adjuvant hormonal management.
* Patient must be willing to undergo a duct lavage.
* Patient must sign an Informed Consent.

Exclusion Criteria:

* None.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients receiving standard Arimidex treatment.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2002-11; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Antiproliferative Effects of Arimidex | Study duration 4 years
  Biomarker modulation study on effects of Armimidex in ductal lavage fluid from evaluable epithelial cells specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org